CLINICAL TRIAL: NCT01149577
Title: Effect of Olanzapine on Sleep Electroencephalogram (EEG) in Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Psychiatry, Ranchi, India (Other)
Responsible Party: S Haque Nizamie, Central Institute of Psychiatry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCHOLZ0003
Record Dates: First submitted 2010-06-18; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia; Sleep
Keywords: Olanzapine; Schizophrenia; Polysomnography; Slow wave sleep
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Schizophrenia patients (Experimental): The study population of 25 schizophrenia patients constituted the active arm of the study.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — 06 weeks treatment with Olanzapine in a flexible dosage schedule.

SUMMARY:
Acute and sub-chronic administration of olanzapine has shown a favourable effect on the sleep disturbances in previously medicated schizophrenia patients with predominantly negative symptoms. The present study will be carried out to clarify the effect of olanzapine on polysomnographic profiles of schizophrenia patients in an acute phase of illness after controlling for the drug effects.

DETAILED DESCRIPTION:
Twenty schizophrenia patients (11 drug naïve and 9 drug free) will be studied over a period of six weeks of olanzapine treatment. Patients will be assessed at the baseline on BPRS, PANSS, CDSS and UKU side effect rating scales and a baseline 40 channels polysomnography will be done. After the initial assessment, patients will put on olanzapine treatment, in flexible dosages based on clinical response, for a period of six weeks when a final assessment on clinical rating scales and polysomnography will be done. The sleep data will be scored manually for staging based on Rechtschaffen and Kales criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients fulfilling International Classification of Diseases-10 Diagnostic Criteria for Research for schizophrenia
2. Aged 18-50 Yrs
3. Drug naïve or drug free (not receiving any psychotropic medication for the past 4 months)
4. Consenting

Exclusion Criteria:

1. Any comorbid psychiatric illness
2. Significant medical or neurological illness
3. History of significant head injury, epilepsy
4. Substance use in the past 4 months excluding nicotine and caffeine
5. Presence of a primary sleep disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Sleep EEG | 06 weeks
  Changes in Sleep EEG parameters like Total sleep time, total sleep period, sleep efficiency, sleep latency, stage shifts, stage 1 shifts, stage 1 parameters, stage 2 parameters, stage 3 parameters, stage 4 parameters, rapid eye movement (REM) parameters.

SECONDARY OUTCOMES:
Psychopathology | 06 weeks
  Changes in psychopathological scores as measured by Brief Psychiatric Rating Scale (BPRS) and Positive and Negative Syndrome Scale (PANSS).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Zia Ul Haq Katshu, DPM, Principal Investigator — Central Institute of Psychiatry
Locations (1):
- Central Institute of Psychiatry, Ranchi, Jharkhand, India